CLINICAL TRIAL: NCT06670599
Title: Neutrophil-to-Lymphocyte and Platelet-to-lymphocyte Ratios as a Predictor Factors for Chronic Kidney Disease Progression
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Said Ashamallah Said, Doctor, Assiut University
Other Study IDs: NLR & PLR in CKD.
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: CKD
Keywords: NLR & PLR in CKD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we aim to investigate whether NLR and PLR levels are associated with decline of kidney function in patients with CKD.

DETAILED DESCRIPTION:
Chronic inflammation is closely associated with various chronic diseases, such as diabetes mellitus, cardiovascular disease, and chronic kidney disease (CKD) (1). Patients with CKD tend to have elevated levels of inflammatory mediators, including high-sensitivity C-reactive protein (hs-CRP), tumor necrosis factor alpha (TNF alpha), and interleukin (IL)-6 (2).These mediators stimulate inflammatory pathway, leading to glomerular hypertension, tubulointerstitial fibrosis, kidney scarring, and, finally, CKD progression and increased cardiovascular events (3,4). Therefore, it is important to evaluate and decrease the extent of chronic inflammation in patients with CKD. Patients with CKD have higher levels of proinflammatory cytokines, but it remains unclear which biomarker is the best indicator of inflammation in patients with CKD.

The neutrophil-to-lymphocyte ratio (NLR), obtained by dividing the absolute number of neutrophils to the lymphocyte count, is increasingly studied as a new inflammatory marker. An elevated NLR has recently been reported to be an independent predictor of mortality in patients with cardiovascular disease or cancer [5-8]. As CKD is a chronic inflammatory disease, high NLR can predict CKD progression, cardiovascular disease and cancer. However, significantly few studies have investigated the association between high NLR and CKD progression [9-12].

Platelet-to-lymphocyte ratio (PLR) has recently been recognized as a novel inflammatory marker and has been shown to be associated with the prognosis in CKD patients [13].

In 2012, Kidney Disease: Improving Global Outcome (KDIGO) classified CKD in six categories by GFR estimation (in mL/min/1.73 m2).

ELIGIBILITY:
Inclusion Criteria:

* 200 Patients diagnosed with CKD and their age range between 18-65 years old who will be admitted at AUH.

Exclusion Criteria:

1. Pediatric patients aged below< 18 or elderly patients aged above 65.
2. Pregnant females.
3. Patients with Diabetes Mellitus.
4. Acute kidney injury (AKI).
5. Patients with current infections.
6. Patients who have any type of malignancy.
7. Patients who have any type of multi-organ failure.
8. CKD patients on dialysis

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prevalence of Chronic Kidney disease (CKD) in 2017 was 7.1 million individuals globally and in Egypt was 106 patients per 1000 population estimated by (GBD) the Global Burden of Disease.
  In September 2021, about 10% of adult population is estimated to have CKD in the world, but the prevalence is higher in Egypt accounted for about 15-20% of adults.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between NLR, PLR and severity of CKD. | Baseline
  Correlation between NLR, PLR and severity of CKD.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gan W, Guan Q, Hu X, Zeng X, Shao D, Xu L, Xiao W, Mao H, Chen W. The association between platelet-lymphocyte ratio and the risk of all-cause mortality in chronic kidney disease: a systematic review and meta-analysis. Int Urol Nephrol. 2022 Nov;54(11):2959-2967. doi: 10.1007/s11255-022-03234-0. Epub 2022 May 17. PMID 35581444
- [Result] Altunoren O, Akkus G, Sezal DT, Ciftcioglu M, Guzel FB, Isiktas S, Torun GI, Uyan M, Sokmen MF, Sevim HA, Sarisik FN, Senel ME, Erken E, Gungor O. Does neutrophyl to lymphocyte ratio really predict chronic kidney disease progression? Int Urol Nephrol. 2019 Jan;51(1):129-137. doi: 10.1007/s11255-018-1994-7. Epub 2018 Oct 1. PMID 30276600
- [Result] Navarro JF, Milena FJ, Mora C, Leon C, Garcia J. Renal pro-inflammatory cytokine gene expression in diabetic nephropathy: effect of angiotensin-converting enzyme inhibition and pentoxifylline administration. Am J Nephrol. 2006;26(6):562-70. doi: 10.1159/000098004. Epub 2006 Dec 13. PMID 17167242
- [Result] Turkmen K, Guney I, Yerlikaya FH, Tonbul HZ. The relationship between neutrophil-to-lymphocyte ratio and inflammation in end-stage renal disease patients. Ren Fail. 2012;34(2):155-9. doi: 10.3109/0886022X.2011.641514. Epub 2011 Dec 16. PMID 22172001
- [Result] Manabe I. Chronic inflammation links cardiovascular, metabolic and renal diseases. Circ J. 2011;75(12):2739-48. doi: 10.1253/circj.cj-11-1184. Epub 2011 Nov 8. PMID 22067929